CLINICAL TRIAL: NCT02607124
Title: A Phase I/II Study of Ribociclib, a CDK4/6 Inhibitor, Following Radiation Therapy in Children With Newly Diagnosed Non-biopsied Diffuse Pontine Gliomas (DIPG) and RB+ Biopsied DIPG and High Grade Gliomas (HGG)
Brief Title: A Phase I/II Study of Ribociclib,a CDK4/6 Inhibitor, Following Radiation Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A competing trial was opened for patient population with combination of ribociclib and everolimus.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011XUS17T
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma; Bithalamic High Grade Glioma
Keywords: DIPG
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RB+ High Grade Glioma (Experimental): Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 600mg daily (DIPG); <21 yrs of age 350 mg/m2/day)
  Interventions: Drug: Ribociclib
- Non-Biopsied Diffuse Instrinsic Pontine Glioma (Experimental): Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 600mg daily (DIPG); <21 yrs of age 350 mg/m2/day)
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib
  Other Names: LEE011

SUMMARY:
In this research study the investigators want to learn more about the effects, both good and bad, when the study drug Ribociclib is given after radiation therapy.

The investigators are asking people to be in this research study that have been newly diagnosed with a high grade glioma, and the tumor has been screened for the Rb1 protein, and have recently finished radiation therapy. Patients with a DIPG or a Bi-thalamic high grade glioma do not need to have tumor tissue screened for the Rb1 protein but do need to have finished radiation therapy.

Tumor cells grow and divide quickly. In normal cells, there are proteins called cyclin-dependent kinases (CDK 4 and 6) that control cell division. Another protein Rb1 also controls cell division and works to stop cells from dividing so they do not become cancer cells. But in cancer, the CDK 4 and 6 proteins are out of control making the cells divide and grow quickly. The study drug, ribociclib stops the CDK 4 and 6 proteins. When the CDK 4 and 6 proteins are stopped, the normal Rb1 protein can now work to slow cell growth. For patients with HGG, to be in this study tumor tissue must have a normal Rb1 protein. The researchers think that if the study drug is given soon after radiation therapy, it may help improve the effect of the radiation in stopping the tumor from growing.

The study drug, Ribociclib is considered investigational as it has not yet been approved by the United States Food and Drug Administration. The study drug has been tested in children and adults with cancer in prior research studies.

DETAILED DESCRIPTION:
Ribociclib has shown an acceptable toxicity profile in adults and pediatrics. Available data suggests that over 70% of DIPG patient have an intact RB and 90% HGG patients have expression of RB, therefore CDK4/6 inhibition is a suitable target. Given the dismal prognosis for children with DIPG and HGG, it is appropriate to evaluate the long term feasibility and early efficacy of Ribociclib following radiation therapy in patients with RB+ tumors. The aim of the upfront biopsy molecular studies proposed is to identify subgroups of patients who will benefit from the use of checkpoint inhibitors in the setting of intact RB pathway. This study will play a major role in moving the field of DIPG/HGG research forward as the investigators intend to reveal feasibility of upfront stereotactic biopsy and specific pathway directed therapy following radiation therapy with the ultimate goal to add additional targeted therapy in combination with Ribociclib resulting in improving the outcome for patients diagnosed with these fatal tumors.

The current proposal will be a novel pediatric study to obtain biopsy in DIPG prior to therapy and administer molecularly targeted therapy following radiation therapy in children with newly diagnosed DIPG and HGG. In this study, the investigators will assess the assess long-term feasibility and early efficacy of Ribociclib administered daily for 3 weeks and off one week every 28 days following radiation therapy for at least 6 courses and up to 12 courses in patients with newly-diagnosed non-biopsied DIPG and RB+ biopsied DIPG and HGG. Moreover, the investigators will approach this devastating disease with a multi-disciplinary team and evaluate the quality of life and functional outcome resulting in effective interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * Patients must be ≥ 12 months of age and ≤ 30 years of age at the time of study entry for patients diagnosed with DIPG.
  * Patients must be ≥ 12 months of age and ≤ 21 years of age at the time of study entry for patients diagnosed with HGG.
* RB status

  * Diagnostic stereotactic biopsy: Patients diagnosed with DIPG may choose to have a stereotactic biopsy prior to starting radiation therapy.
  * Toxicities related to biopsy must have resolved prior to proceeding with radiation therapy.
  * Screening for Rb applies to all patients with available tissue except for patients diagnosed with DIPG and bi-thalamic tumors.
  * If resection occurred at an outside institution, eligibility and treatment MRI evaluations in addition to Rb testing must be completed at CCHMC.
* Tumor

  * Diffuse Intrinsic Pontine Glioma (DIPG) Patients with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined on neuroimaging as tumors with a pontine epicenter and diffuse intrinsic involvement of the pons, are eligible without histologic confirmation.
  * Patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors are biopsied and proven to have + RB and be the following according to the 2016 World Health Organization classification of tumors of the central nervous system: an anaplastic astrocytoma (IDH mutant, IDH wildtype, or NOS), glioblastoma (IDH mutant, IDH wildtype or NOS), diffuse midline glioma, H3 K27M mutant or H3 K27M negative, diffuse astrocytoma (IDH mutant, IDH wildtype or NOS).
  * Note: Patients with juvenile pilocytic astrocytoma, pilomyxoid astrocytoma, pleomorphic xanthoastrocytoma with or without anaplasia, gangliogliomas, or other mixed gliomas without anaplasia are not eligible.
  * Patients with diffuse intrinsic brain stem glioma (DIPG) can be enrolled without the need for available tumor tissue for RB protein status confirmation.
  * Bi-thalamic tumors, biopsied and noted to have intact RB. Bi-thalamic tumors that are not biopsied will be eligible to enroll on the DIPG/bi-thalamic non-biopsied arm.
  * High-grade Glioma (HGG)
  * Patients must have had histologically verified the following according to the 2016 World Health Organization classification of tumors of the central nervous system: anaplastic astrocytoma (IDH mutant, IDH wildtype, or NOS), glioblastoma multiforme (IDH mutant, IDH wildtype, or NOS), diffuse astrocytoma (IDH mutant, IDH wildtype or NOS)
  * AND RB positive noted on immunohistochemistry.
  * Patients with primary spinal cord tumors are eligible. Patients with multi-focal disease within the cerebrum are eligible.
  * Patients with a diagnosis of oligodendroglioma or oligoastrocytoma are not eligible.
* Performance Status

  • Karnofsky > 50 % for patients >16 years of age or Lansky > 50 for patients < 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy

  • Patients must have not received any prior therapy other than surgery, radiation and/or steroids.
* Radiation therapy requirements

  * Patients diagnosed with DIPG: any variances in the radiotherapy dose within 10% of the current standard dose (54 Gy) will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment
  * Patients diagnosed with HGG: any variances in the radiotherapy dose within 10% of the current standard dose (59.4 Gy) will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.
  * Patients diagnosed with primary spinal tumors any variances in the radiotherapy dose within 10% of the current standard dose (54 Gy) will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.
  * Timing of Radiation - radiation therapy must begin no later than 30 days after the date of radiographic diagnosis or definitive surgery, whichever is the later date.
* Organ Function

  * Patients must have normal organ and marrow function documented within 7 days of study enrollment as defined below:
  * Absolute neutrophil count ≥ 1000mm3
  * Platelets ≥ 75,000/mm3 (unsupported for 7 days)
  * Hemoglobin ≥ 9g/dl (unsupported) for 7 days
  * Total bilirubin ≤ 3 times upper limit of normal (ULN) for age
  * ALT (SGPT) ≤ 2.5 X ULN for age
  * Albumin ≥ 2 g/dl
  * Creatinine clearance or radioisotope GFR ≥ 70mL/min/1.73m2 or serum creatinine based on age/gender.
* Pregnancy Status Female patients of childbearing potential, must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test.
* Pregnancy Prevention Patients of childbearing or child fathering potential must use a highly effective method of contraception throughout the study while taking the drug and for 21 days after stopping treatment
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Informed Consent Signed informed consent according to institutional guidelines must be obtained. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Concurrent Illness Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results.
* Inability to Participate Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.
* Received a radiosensitizer or any additional adjuvant therapy during radiation therapy.
* Patients with disseminated disease to the spine are not eligible, and MRI of spine must be performed prior to enrollment if the treating physician suspects disseminated disease.
* Seizures Patients who are currently receiving enzyme inducing anti-epileptic drugs that are known strong inducers or inhibitors of CYP3A4/5 (EIAEDs). Patients with a history of seizures and maintained on an anti-epileptic drug that is not a strong inducers or inhibitor of CYP3A4/5 are eligible.
* Patient has a known hypersensitivity to Ribociclib or any of its excipients.
* Clinically significant active cardiac disease, uncontrolled heart disease and/or history of cardiac dysfunction including any of the following

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Patient has a Left Ventricular Ejection Fraction (LVEF) < 50 % as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
  * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
  * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
  * Hypertension defined below:
  * Patients 2-17 years of age must have a blood pressure that is ≤ 95th percentile for age, height and gender at the time of enrollment.
  * Patients who are ≥ 18 years of age must have a systolic blood pressure that is > 160 or diastolic < 90 mm of Hg at the time of enrollment
  * Note: If a BP reading prior to enrollment is above the 95th percentile for age, height and gender, it is to be rechecked and documented to be ≤ 95th percentile for age, height and gender prior to patient enrollment.
* Inability to determine the QTcF interval on the ECG (i.e. unreadable or not interpretable) or QTcF > 450 msec (using Fridericia's correction). All as determined by screening ECG (using the mean QTcF of triplicate ECGs)
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug Ribociclib:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pomelos, star-fruit, and Seville oranges
  * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Medications that have a known risk to prolong the QT interval or induce Torsades de Pointes
  * Herbal preparations/medications, dietary supplements.
* Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed
* Patient has a history of non-compliance to medical regimen.
* Known need for major surgery within 14 days of the first dose of Ribociclib. Gastrostomy, insertion of a G tube, Ventriculo-peritoneal shunt, endoscopic ventriculostomy and central venous access are NOT considered major surgery.

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariko DeWire, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] DeWire M, Fuller C, Hummel TR, Chow LML, Salloum R, de Blank P, Pater L, Lawson S, Zhu X, Dexheimer P, Carle AC, Kumar SS, Drissi R, Stevenson CB, Lane A, Breneman J, Witte D, Jones BV, Leach JL, Fouladi M. A phase I/II study of ribociclib following radiation therapy in children with newly diagnosed diffuse intrinsic pontine glioma (DIPG). J Neurooncol. 2020 Sep;149(3):511-522. doi: 10.1007/s11060-020-03641-2. Epub 2020 Oct 9. PMID 33034839
- [Derived] Gilligan LA, DeWire-Schottmiller MD, Fouladi M, DeBlank P, Leach JL. Tumor Response Assessment in Diffuse Intrinsic Pontine Glioma: Comparison of Semiautomated Volumetric, Semiautomated Linear, and Manual Linear Tumor Measurement Strategies. AJNR Am J Neuroradiol. 2020 May;41(5):866-873. doi: 10.3174/ajnr.A6555. Epub 2020 Apr 30. PMID 32354716

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Biopsied Diffuse Instrinsic Pontine Glioma/Diffuse Midline Glioma: Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 600mg daily (DIPG); <21 yrs of age 350 mg/m2/day)
Period: Overall Study
Arm/Group | Non-Biopsied Diffuse Instrinsic Pontine Glioma/Diffuse Midline Glioma
Started | 10 (11 participants were enrolled however 1 participant withdrew before starting study treatment.)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Demographics for participants are combined for enrolled participants stratified by diagnosis. Intervention was identical for all diagnoses.
Groups:
- Diffuse Instrinsic Pontine Glioma and Diffuse Midline Glioma: Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 600mg daily (DIPG); <21 yrs of age 350 mg/m2/day)
  Baseline characteristics data are collected irrespective of Arm/Group and cannot be reported separately.
Arm/Group | Diffuse Instrinsic Pontine Glioma and Diffuse Midline Glioma
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: One enrolled participant was ineligible for study treatment and removed from trial therefore deemed inevaluable.
  Participants
    <=18 years | 9
    Between 18 and 65 years | 1
    >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 7.5 [3.8 to 20.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Primary feasibility endpoint is the number of individual toxicities and incidence of significant delays
Time Frame: 6 months
Population: Number of participants receiving investigational agent.
Measure: Number; unit: adverse event
Groups:
- RB+ High Grade Glioma; Non-Biopsied Diffuse Instrinsic Pontine Glioma: Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 600mg daily (DIPG); <21 yrs of age 350 mg/m2/day)
  Ribociclib
Arm/Group | RB+ High Grade Glioma | Non-Biopsied Diffuse Instrinsic Pontine Glioma
Number analyzed (Participants) | 1 | 9
adverse event | 9 | 144

2. Primary Outcome: Number of Patients Alive at One Year
Time Frame: 1 year
Population: Number of enrolled and evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | RB+ High Grade Glioma | Non-Biopsied Diffuse Instrinsic Pontine Glioma
Number analyzed (Participants) | 1 | 9
Participants | 0 | 8

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events grades 1 and 2 that are at least possibly related to ribociclib and all adverse events grades 3 and higher regardless of attribution during study treatment were recorded for the purposes of safety monitoring.
  There were no serious adverse events attributable to study treatment.
Groups:
- Diffuse Intrinsic Pontine Glioma and High Grade Glioma: Ribociclib administered orally; daily on days 1-21 each 28 day cycle; dose calculation age dependent (>21 yrs of age 600mg daily (DIPG); <21 yrs of age 350 mg/m2/day)
Arm/Group | Diffuse Intrinsic Pontine Glioma and High Grade Glioma
All-Cause Mortality (participants affected / at risk) | 10/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Intrinsic Pontine Glioma and High Grade Glioma (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1
Accessory nerve disorder (Nervous system disorders) | 1
agitation (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysarthria (Nervous system disorders) | 1
Gait Disturbance (General disorders) | 1
hallucination (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection-Other (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Nervous system disorders - Other, specify (hemiparesis) (Nervous system disorders) | 1
Non Cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (tachypnea) (Respiratory, thoracic and mediastinal disorders) | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Intrinsic Pontine Glioma and High Grade Glioma (N=10)
Anemia (Blood and lymphatic system disorders) | 6
Vomiting (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastroesophageal reflux diease (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Gait Disturbance (General disorders) | 1
Pain (General disorders) | 1
Edema limbs (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Creatinine Increased (Investigations) | 10
Ejection fraction decreased (Investigations) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 10
Neutrophil Count Decreased (Investigations) | 10
Platelet Count Decreased (Investigations) | 5
Weight Gain (Investigations) | 2
Weight Loss (Investigations) | 2
White Blood Cell Decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Osteonecrosis - hip) (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Other - Rash (Skin and subcutaneous tissue disorders) | 1
Other - petechial rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT02607124/Prot_SAP_000.pdf